CLINICAL TRIAL: NCT06107569
Title: Randomized Controlled Clinical Study of Treatment of Clostridioides Difficile Infection Comparing Fecal Microbiota Transplantation With Antibiotic Treatment
Brief Title: Treatment of CDI and Recurrence With Fecal Microbiota Transplant Using Promicrobioma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitario Evangelico de Curitiba (Other)
Responsible Party: Principal Investigator, Felipe Francisco Bondan Tuon, Principal Investigator, Hospital Universitario Evangelico de Curitiba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDItransplant
Record Dates: First submitted 2023-10-13; First posted 2023-10-30 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Clostridium Difficile Infections
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Promicrobioma (Experimental): MIcrobiote tranplant
  Interventions: Other: Fecal microbiota transplant (Promicrobioma)
- Antibiotic (metronidazole or vancomycin) (Active Comparator): Antibiotic commonly used for treatment of CDI, including oral vancomycin or metronidazol)
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Other: Fecal microbiota transplant (Promicrobioma) — Fecal microbiota transplant with Promicrobioma (freeze-dried isolated microbiota)
  Arms: Promicrobioma
Drug: Antibiotic — Antibiotics for Clostridioides infection (oral vancomycin) or association of intravenous metronidazol for severe cases.
  Arms: Antibiotic (metronidazole or vancomycin)

SUMMARY:
The increasing inappropriate use of antimicrobials, in addition to increasing selective pressure and inducing environmental resistance, is also a risk factor for the development of Clostridioides difficile infection (CDI). The intestinal microbiota is mainly composed of the phyla Firmicutes, Bacteroidetes, Acinobacteria, Proteobacteria, Fusobacteria and Verrucomicrobia, and more than 90% of the phylum Firmicutes is composed of Clostridium spp. (two). The inappropriate use of antimicrobials initiates a process of dysregulation of the microbiome, called dysbiosis, and it is from the selection of genera and species of bacteria that will dominate the intestine that pseudomembranous colitis can set in with an increased burden of Clostridioides difficile, a gram positive, anaerobic, spore-forming, that produces two enterotoxins, toxin A and toxin.

DETAILED DESCRIPTION:
INTRODUCTION

The increasing inappropriate use of antimicrobials, in addition to increasing selective pressure and inducing environmental resistance, is also a risk factor for the development of Clostridioides difficile infection (CDI). The intestinal microbiota is mainly composed of the phyla Firmicutes, Bacteroidetes, Acinobacteria, Proteobacteria, Fusobacteria and Verrucomicrobia, and more than 90% of the phylum Firmicutes is composed of Clostridium spp. (two). The inappropriate use of antimicrobials initiates a process of dysregulation of the microbiome, called dysbiosis, and it is from the selection of genera and species of bacteria that will dominate the intestine that pseudomembranous colitis can set in with an increased burden of Clostridioides difficile, a gram positive, anaerobic, spore-forming, that produces two enterotoxins, toxin A and toxin.

Currently, pseudomembranous colitis has few treatment options: the main one is fidaxomicin, unavailable in Brazil, and other alternatives are vancomycin and metronidazole. However, refractoriness to alternative treatments may occur, with fecal transplantation also being an alternative. Additionally, fecal transplantation is often associated with better outcomes than drug alternatives, reaching more than 90% clinical success.

Fecal microbiota transplantation (FMT) can occur through different routes, for example, via nasoenteral tube, colonoscopy, oral capsules or enemas, with colonoscopy or capsules normally being apparently more effective than enemas and nasoenteral tubes. Furthermore, the preparation of stool samples can be either fresh or frozen, which do not influence the effectiveness of the treatment. Since 2020, the PUCPR Fecal Microbiota Bank has been carrying out validation studies of a product, PROMICROBIOMA, composed of freeze-dried human fecal microbiota, which has already tested its safety in a phase 1 study on consecutive patients in a convenience sample. To evaluate the effectiveness of the product, it is important to carry out a controlled and randomized clinical study comparing it with antimicrobial therapy.

HYPOTHESIS H0 - PROMICROBIOMA is equal to antibiotic treatment in primary or recurrent CDI H1 - PROMICROBIOME is superior to antibiotic treatment in primary or recurrent CDI H2 - PROMICROBIOME is inferior to antibiotic treatment in primary or recurrent CDI

MAIN GOAL

To evaluate the clinical outcome of patients with primary or recurrent CDI using PROMICROBIOMA compared to antimicrobial therapy.

METHODS

Study design

This is a randomized, controlled clinical study of patients with primary or recurrent CDI.

ELIGIBILITY:
The inclusion criteria are:

1. Over 18 years old;
2. Hospitalized patients;
3. Clinical and laboratory diagnosis of CDI;
4. Signing the informed consent form
5. For primary CDI, use of antibiotics for less than 72 hours; and for recurrent CDI, previous confirmed CDI with clinical response to antibiotic treatment and CDI recurrence within 8 weeks.

The exclusion criteria are:

1. Pregnant patients
2. Severe form of CDI requiring surgery
3. Impossibility of performing the colonoscopy procedure or using a nasoenteral tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate | 8 weeks
  Clinical cure is defined as absence of diarrhea, abdominal pain, clinical signs of infection (fever).